CLINICAL TRIAL: NCT04266678
Title: Changes to Muscle Quality and Sarcopenia Status After Short-Term Resistance Training in Older Adults
Brief Title: Short-Term Resistance Training in Older Adults
Acronym: OART
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Kansas (Other)
Responsible Party: Principal Investigator, Ashley Herda, Assistant Professor, University of Kansas
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: STUDY00143495
Record Dates: First submitted 2020-02-10; First posted 2020-02-12 (Actual); Last update posted 2021-04-28 (Actual); Status verified 2021-04

CONDITIONS: Sarcopenia; Muscle Quality
Keywords: muscular strength; functional capacity; resistance exercise
MeSH Terms: conditions — Sarcopenia

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Elastic band resistance training (Experimental): Resistance training with elastic resistance bands two days per week for 6-weeks.
  Interventions: Behavioral: Resistance exercise program
- Dumbbell resistance training (Active Comparator): Resistance training with dumbbell weights two days per week for 6-weeks.
  Interventions: Behavioral: Resistance exercise program
- Non-exercise Control (No Intervention): Education and guidance for exercise recommendations in older adults but no active training sessions.

INTERVENTIONS:
Behavioral: Resistance exercise program — Exercise sessions with exercise science professional. Target hypertrophy repetition range and progressive resistance exercise.
  Other Names: control-no exercise
  Arms: Dumbbell resistance training; Elastic band resistance training

SUMMARY:
The purpose of this study will be to evaluate whether dumbbell resistance training (DBRT) or elastic band resistance training (EBRT) is beneficial in older adults whom may be classified as sarcopenic based on the collective operational definition and older adults that do not meet the criteria to be considered sarcopenic compared to non-exercise controls of these populations after sarcopenia criteria have been established. As well as identify if resistance exercise will improve muscle quality in older adults, considering how muscle quality relates to sarcopenia status. Specific Aim 1 will determine if short-term resistance training will alter muscle quality or sarcopenia status in older adults compared to non-exercise controls. The study team will instruct and supervise adults aged 55-85 in structured, periodized EBRT or DBRT for 6 weeks. After the training, muscle quality and sarcopenia status will be re-evaluated. It is hypothesized that both types of training (EBRT and DBRT) will improve the sarcopenia status of older adults engaging in resistance training and if sarcopenic, their classification may change to non-sarcopenic. A secondary hypothesis is that EBRT will be more beneficial than DBRT, resulting in greater changes in body composition, strength, and functional movements. It is also hypothesized that muscle quality, as an index of relative strength, will improve after 6 weeks of resistance training with either dumbbells or elastic bands and that there is a strong negative linear relationship between severity of sarcopenia and muscle quality. Specific Aim 2 will evaluate the prevalence of sarcopenia in older adults using previously-identified equations and cut-off values and to subsequently generate a new index to include functional muscle mass and performance to identify sarcopenic individuals. This will be completed using muscle mass estimations from dual-energy x-ray absorptiometry (DEXA), bioelectrical impedance analysis (BIA), functional performance measures, and structural composition. It is hypothesized that DEXA and BIA will provide accurate estimates of appendicular lean mass (ALM), and functional performance (handgrip strength and gait speed) will be significant contributors to a predictive equation of a muscle quality index for men and women.

DETAILED DESCRIPTION:
It is well known that as adults age, a proportion of lean body mass is reduced if not lost, specifically fast twitch (FT or Type II) fibers, and subsequently, strength and power is diminished. The age-related loss of muscle mass and function is referred to as sarcopenia. Reduction of muscle mass plays a direct role in the loss of function, and potentially, the ability to complete activities of daily living. It is also highly related to an increase in incidence of falls and onset of many other comorbidities resulting in changes in quality of life (QOL). Copeland et al. recently reported that strength training will benefit all adults, regardless of their functional level, based on a self-report survey of nearly 10,000 adults aged 60 years and older. Aside from diagnosing sarcopenia in individuals using pre-identified criteria (and doing so accurately), it is of the utmost importance to implement resistance exercise programs in populations of older adults that can directly combat the decline in type II fiber size, maintain aerobic fitness, aid in maintaining or reducing total body fat, minimize the prevalence of sarcopenia, and ultimately improve QOL. Targeted interventions that include dumbbell and elastic band resistance training (both considered free-movement) and progressive programming schemes have been reported to enhance muscle size, strength, and quality, functional mobility, and confidence in older adults, in turn, reducing percent body fat, risk of falls, and incidence of comorbidities that are often coupled with senescence. Recently, Calatayud et al. reported similar improvements in strength and muscle activation (electromyographic [EMG] amplitude) between free weight (bench press) and resistance band (band push-up) exercises, suggesting either mode of resistance exercise would be beneficial. Furthermore, use of resistance bands for chest flys and reverse flys were validated to be comparable with conventional free weights. There are several exercises that can be duplicated using either modality. However, the challenge is the vertical plane for free weights, as free weights only provide resistance against gravity and exercise movements, more specifically, body position, need to be modified in order to perform the resisted movement. Some older adults tend to have balance impairments and thus adjusting their body position to perform (dumbbell) resisted exercise may not be ideal, specifically if they may have a greater risk for falls as suggested by sarcopenia status (i.e. reduced muscle mass and gait speed or strength). Therefore the purpose of this study will be to evaluate whether dumbbell resistance training (DBRT) or elastic band resistance training (EBRT) is beneficial in older adults whom may be classified as sarcopenic based on the collective operational definition and older adults that do not meet the criteria to be considered sarcopenic compared to non-exercise controls of these populations after sarcopenia criteria have been established. As well as identify if resistance exercise will improve muscle quality in older adults, considering how muscle quality relates to sarcopenia status.

ELIGIBILITY:
Inclusion Criteria:

* Subject has provided written and dated informed consent to participate in the study.
* Subject is a male or female between 55 and 85 years of age, inclusive.
* Subject is in good health as determined by a health history questionnaire and has been provided clearance from their personal physician.
* Subject is untrained in resistance and aerobic exercise (does not participate in structured physical activity, including walking, more than 3 times per week).

Exclusion Criteria:

* Subject has a history of alcohol or other drug abuse in the past year.
* Subject has a history or current presence of congestive heart failure, or any other form of cardiovascular disease that might put the subject at risk.
* Subject has a significant history or current presence of untreated bleeding disorder, diabetes mellitus, high blood pressure (BP) [systolic BP> 140 and/or diastolic BP> 90], thyroid disease, tachyarrhythmia, heart disease, kidney disease, or liver disease.
* Subject currently suffers from a sleep disorder and/or has a known history of (or is currently being treated for) clinical depression, eating disorder(s) or any other psychiatric condition(s) that might put the subject at risk and/or confound the results of the study.
* Subject has a history of orthopedic injury or surgery within the last year that may prevent them from completing the study procedures.
* Subject has arthritis of the hand which could impair his/her ability to grip a dynamometer.
* Subject has severe arthritis defined as grade 3 or higher as diagnosed by a physician.
* No history of CT scans (computed tomography), PET and nuclear medicine studies, or fluoroscopic procedures within the past year. Nuclear medicine imaging studies use agents that will interfere with the DXA whole body scan.
* No implants, hardware, devices, or other foreign material in the measurement area. These devices will make whole body measurements difficult to interpret when the devices or implants are located within the scan field.

Ages: 55 Years to 85 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 73 (Actual)
Dates: Start 2019-04-09 (Actual); Primary Completion 2020-03-16 (Actual); Study Completion 2020-10-30 (Actual)

PRIMARY OUTCOMES:
Muscle mass | 6-weeks
  Quantity of upper and lower body muscle mass with DXA (in kg)
Upper and lower body strength | 6-weeks
  Maximal amount of weight lifted in 5 repetitions for bench press and leg press

SECONDARY OUTCOMES:
Fat mass | 6-weeks
  Quantity of fat assessed by DXA
Short Physical Performance Battery (SPPB) | 6-weeks
  gait speed and balance tests
Handgrip Strength | 6-weeks
  maximal dominant hand handgrip strength (in kg)

CONTACTS AND LOCATIONS:
Overall Officials: Ashley A Herda, PhD, Principal Investigator — University of Kansas
Locations (1):
- University of Kansas-Edwards Campus; Exercise and Human Performance Laboratory, Overland Park, Kansas, United States

IPD SHARING:
Plan to Share IPD: Undecided
If required for publication, IPD will be made available through an Institution-supported database server.

REFERENCES:
- [Background] Baumgartner RN, Wayne SJ, Waters DL, Janssen I, Gallagher D, Morley JE. Sarcopenic obesity predicts instrumental activities of daily living disability in the elderly. Obes Res. 2004 Dec;12(12):1995-2004. doi: 10.1038/oby.2004.250. PMID 15687401
- [Background] Bergquist R, Iversen VM, Mork PJ, Fimland MS. Muscle Activity in Upper-Body Single-Joint Resistance Exercises with Elastic Resistance Bands vs. Free Weights. J Hum Kinet. 2018 Mar 23;61:5-13. doi: 10.1515/hukin-2017-0137. eCollection 2018 Mar. PMID 29599855
- [Background] Calatayud J, Borreani S, Colado JC, Martin F, Rogers ME. Muscle activity levels in upper-body push exercises with different loads and stability conditions. Phys Sportsmed. 2014 Nov;42(4):106-19. doi: 10.3810/psm.2014.11.2097. PMID 25419894
- [Background] Copeland JL, Good J, Dogra S. Strength training is associated with better functional fitness and perceived healthy aging among physically active older adults: a cross-sectional analysis of the Canadian Longitudinal Study on Aging. Aging Clin Exp Res. 2019 Sep;31(9):1257-1263. doi: 10.1007/s40520-018-1079-6. Epub 2018 Nov 27. PMID 30484254
- [Background] Nilwik R, Snijders T, Leenders M, Groen BB, van Kranenburg J, Verdijk LB, van Loon LJ. The decline in skeletal muscle mass with aging is mainly attributed to a reduction in type II muscle fiber size. Exp Gerontol. 2013 May;48(5):492-8. doi: 10.1016/j.exger.2013.02.012. Epub 2013 Feb 17. PMID 23425621
- [Background] Schrack JA, Zipunnikov V, Simonsick EM, Studenski S, Ferrucci L. Rising Energetic Cost of Walking Predicts Gait Speed Decline With Aging. J Gerontol A Biol Sci Med Sci. 2016 Jul;71(7):947-53. doi: 10.1093/gerona/glw002. Epub 2016 Feb 5. PMID 26850913
- [Background] Skelton DA, Greig CA, Davies JM, Young A. Strength, power and related functional ability of healthy people aged 65-89 years. Age Ageing. 1994 Sep;23(5):371-7. doi: 10.1093/ageing/23.5.371. PMID 7825481
- [Background] Snijders T, Nederveen JP, Bell KE, Lau SW, Mazara N, Kumbhare DA, Phillips SM, Parise G. Prolonged exercise training improves the acute type II muscle fibre satellite cell response in healthy older men. J Physiol. 2019 Jan;597(1):105-119. doi: 10.1113/JP276260. Epub 2018 Nov 24. PMID 30370532
- [Background] Yoshiko A, Tomita A, Ando R, Ogawa M, Kondo S, Saito A, Tanaka NI, Koike T, Oshida Y, Akima H. Effects of 10-week walking and walking with home-based resistance training on muscle quality, muscle size, and physical functional tests in healthy older individuals. Eur Rev Aging Phys Act. 2018 Nov 19;15:13. doi: 10.1186/s11556-018-0201-2. eCollection 2018. PMID 30473735

DOCUMENTS (1):
  • Informed Consent Form (2020-02-07): https://cdn.clinicaltrials.gov/large-docs/78/NCT04266678/ICF_000.pdf